CLINICAL TRIAL: NCT05728229
Title: Effetti Della Nutrizione Sulla Fatica Post Stroke
Brief Title: Effects of Nutrition on Post Stroke Fatigue
Acronym: NUTRE-S
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, GIOVANNINI SILVIA, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0033318/22
Record Dates: First submitted 2023-02-04; First posted 2023-02-15 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-12

CONDITIONS: Fatigue; Stroke
Keywords: Stroke; Fatigue; Older Adults; Nutrition
MeSH Terms: conditions — Fatigue; Stroke

STUDY DESIGN:
Intervention Model Description: Interventional randomized controlled pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (GS) (Experimental): GS patients, in addition to the pharmacological therapy foreseen by the clinical conditions, will take 1 sachet a day of SiderAl® Med, a food for special purposes, for 28 days. GS patients will take the food for special purposes during hospitalization (between T0 and T1) and during the 1 month of returning home (between T1 and T2). During the second month of returning home (between T2 and T3), GS patients will no longer take the food for special purposes.
  Interventions: Drug: Supplement with SiderAl® Med
- Control Group (GC) (No Intervention): The patients of the GC, on the other hand, will continue to take the drug as required by their clinical conditions and will not take the SiderAL® Med food for special purposes, but will only be observed and evaluated at the various time-points foreseen by the study.

INTERVENTIONS:
Drug: Supplement with SiderAl® Med — Nutritional supplementation with special purpose food
  Other Names: SiderAl® Med
  Arms: Experimental Group (GS)

SUMMARY:
Fatigue, which is commonly defined as a feeling of tiredness during or after usual activities, or a feeling of insufficient energy to initiate these activities, is one of the most common secondary conditions among patients presenting with stroke.

Post Stroke Fatigue (PSF) is a multidimensional motor-perceptual, emotional, and cognitive experience characterized by a feeling of early exhaustion with tiredness, lack of energy, and difficulty making efforts, which develops during physical or mental activities, and usually does not improve with rest.

To try to counteract fatigue and its effects on daily life activities, in addition to the known pharmacological approach (Modafinil), the use of vitamins and minerals is known to mitigate, among others, the effects of fatigue. Nutrients provide the energy needed to maintain the body's structural and biochemical integrity. Energy is associated with a feeling of well-being, increased stamina and vitality which often translates into the ability to undertake daily physical or cognitive activities and social relationships, as opposed to fatigue.

A common feature of fatigue is a "sense of energy exhaustion" which can objectively be related to not enough energy. Physical and cognitive tiredness occurs when the continuous demand for energy from the brain and muscles is not met. In humans, dietary macronutrients provide the fuel needed, among other things, to perform physical activity. In fact, mineral salts and vitamins are essential for the production of cellular energy, for the maintenance of brain structures and for allowing the formation of intercellular connections.

When the intake of vitamins and mineral salts is adequate, their biochemical properties translate into normal physiological functions; a lower intake of mineral salts and vitamins is associated with lethargy and physical and cognitive fatigue. However, few studies have evaluated the effect of vitamin and mineral supplementation for the management of physical and cognitive fatigue.

SiderAL® Med is a food for Special Medical Purposes (AFMS), with a complete formulation that contains vitamins, sucrosomial minerals (Iron, Iodine, Magnesium, Zinc and Selenium), copper and algal calcium, with enhanced dosages to meet particular needs nutritional. AFMS are products formulated for the dietary management of patients with proven nutritional needs, for whom modifications to the normal diet are not sufficient.

In some cases, these are subjects with limited, disturbed or altered ability to take, digest, absorb, metabolize or eliminate certain nutrients, in other cases, however, nutritional needs can be determined by specific clinical conditions.

On the basis of scientific evidences, therefore, the aim of the study is to evaluate whether the nutritional supplement with SiderAL® Med improves the symptom of fatigue, motor and cognitive function in patients with stroke outcomes.

DETAILED DESCRIPTION:
Twenty-four patients of both sexes will be recruiteed, evaluated and treated at the Post-Acute Rehabilitation Unit, Fondazione Policlinico Universitario A. Gemelli IRCCS of Rome.

Patients will be divided into two groups by randomization, as specified later. One group (experimental group, GS), in association with the drug therapy already underway, will take the nutritional supplement with SiderAL® Med 1 sachet per day for 28 consecutive days, while another group will continue its clinical and rehabilitation treatment as per the daily routine (control group, GC).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 5 years;
* Patients with ischemic or haemorrhagic stroke outcomes documented through neuroimaging techniques (magnetic resonance or computed tomography);
* Latency from the acute event between 1 and 6 months;
* Cognitive skills that allow you to carry out simple orders and understand the physiotherapist's instructions [assessed through the Token Test (score ≥ 26.5)];
* Ability to walk independently or with little assistance;
* Ability to understand and sign informed consent.

Exclusion Criteria:

* Vitamin D intake greater than 3000 IU/day;
* Therapy with Vitamin K antagonists;
* Conditions causing excess electrolytes in the blood;
* Diagnosis of metabolic mineral storage disorders (eg, hemochromatosis, Wilson);
* Dialysis patients;
* Systemic, neurological, cardiac pathologies that make walking risky or cause motor deficits;
* Oncological pathologies;
* Problems of an orthopedic or postural nature;
* Presence of plantar ulcers;
* Partial or total amputation of segments of the foot;
* Inability to provide informed consent.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-09-29 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | Change from Baseline MFIS at 4, 8 and 16 weeks
  The MFIS is an instrument that provides an assessment of the effects of fatigue in terms of physical, cognitive, and psychosocial functioning. The full-length MFIS consists of 21 items while the abbreviated version has 5 items.
  The MFIS is a structured, self-report questionnaire that the patient can generally complete with little or no intervention from an interviewer. However, patients with visual or upper extremity impairments may need to have the MFIS administered as an interview. Interviewers should be trained in basic interviewing skills and in the use of this instrument.
  The total score for the MFIS is the sum of the scores for the 21 items. Individual subscale scores for physical, cognitive, and psychosocial functioning can also be generated by calculating the sum of specific sets of items.

SECONDARY OUTCOMES:
Fatigue Scale for Motor and Cognitive Function (FSMC) | Change from Baseline FSMC at 4, 8 and 16 weeks
  The FSMC is an assessment of MS-related cognitive and motor fatigue. A Likert-type 5-point scale (ranging from 'does not apply at all' to 'applies completely') produces a score between 1 and 5 for each scored question. Thus minimum value is 20 (no fatigue at all) and maximum value is 100 (severest grade of fatigue). Two subscales (mental and physical fatigue) can be made. Items included in the subscale mental are 1-4-7-8-11-13-15-17-18-20 and items included in the subscale physical are 2-3-5-6-9-10-12-14-16-19.
Berg Balance Scale (BBS) | Change from Baseline BBS at 4, 8 and 16 weeks
  BBS is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.
Short Physical Performance Battery (SPPB) | Change from Baseline SPPB at 4, 8 and 16 weeks
  SPPB is an objective measurement instrument of balance, lower extremity strength, and functional capacity in older adults (>65 years of age). Three domains, which include balance, usual or self-selected gait speed, and lower limb strength, are assessed by a three-stage balance test (feet side-by-side, semitandem, and tandem positions), a 3-m or 4-m gait speed test (time spent to walk the course), and a repetitive chair stand test (five times chair sit-to-stand test), respectively. A 0- to 12-point scale is used to score the sum of the three assessments with higher point values corresponding with greater levels of physical function and lower disability, whereas lower point values correspond with lower levels of physical function and higher disability, respectively.
Motricity Index (MI) | Change from Baseline MI at 4, 8 and 16 weeks
  MI can be used to assess the motor impairment in a patient who has had a stroke.
  Test for each upper limb:
  1. pincer grip
  2. elbow flexion
  3. shoulder abduction
  Test for each lower limb:
  1. ankle dorsiflexion
  2. knee extension
  3. hip flexion
  For the pincer grip:
  0 points, no movement 19 points, grip possible but not against gravity 33 points, normal grip
  For all other items:
  0 points, no movement 14 points, Visible movement but not for the entire joint range or against gravity 19 points, movement possible for the entire joint range against gravity but not against resistance 33 points movement performed with normal force
  Each segment has a total score obtained by adding the value "1" to the score of each individual item. The total score then ranges from 1 (no movement) to 100 (normal movement).
Timed Up and Go Test (TUG) | Change from Baseline TUG at 4, 8 and 16 weeks
  TUG measures in seconds the time it takes a subject to rise from a chair, walk a distance of 3 meters, turn, walk back to the chair and sit down.
  The performance is rated on a scale of 1 to 5 (where 1 is normal and 5 is severely abnormal) according to the observer's perception of the patient's risk of falling.
  The timed part of the test records the mean time (in seconds) from initial getting up to re-seating. Patients are compared with the mean time of adults in their age group, 60 to 69, 70 to 79, and 80 to 99 years of age.
HandGrip Test (HGT) | Change from Baseline HGT at 4, 8 and 16 weeks
  HGT is a test performed with a dynamometer, which goes to assess muscle strength (in kilograms). Starting with the elbow flexed to 90°, the patient must squeeze the dynamometer as hard as they can at one time. Three repeated measurements are taken on each side 20 seconds apart.
  The average of the three assessments is used as the final value.
Ambulation Index (AI) | Change from Baseline AI at 4, 8 and 16 weeks
  AI is a rating scale to assess mobility by evaluating the time and degree of assistance required to walk 8 meters. Scores range from 0 (asymptomatic and fully active) to 10 (bedridden). The patient is asked to walk a marked 8 meters course as quickly and safely as possible. The examiner records the time and type of assistance (e.g., cane, walker, crutches) needed. Although the patient's walking is timed, the time is not used directly but is utilized in conjunction with other factors to rate the patient on an ordinal scale with 11 gradations.
  0 = Asymptomatic; fully active. 10 = Bedridden
Walking handicap scale (WHS) | Change from Baseline WHS at 4, 8 and 16 weeks
  WHS is an assessment tool that allows us to evaluate the quality of walking in the home and social environment through a a scale comprising six categories.
  1 = Physiological walking: walking only as exercise 6 = Unrestricted walking in social settings: independent in all activities, on uneven ground, in crowded places, shows complete independence in public places.
Functional Ambulation Classification (FAC) | Change from Baseline FAC at 4, 8 and 16 weeks
  FAC is a functional walking test that evaluates ambulation ability. This 6-point scale assesses ambulation status by determining how much human support the patient requires when walking, regardless of whether or not they use a personal assistive device.
  To use the FAC, an assessor asks the subject various questions and briefly observes their walking ability to provide a rating from 0 to 5.
  A score of 0 indicates that the patient is a non-functional ambulator (cannot walk); A score of 1, 2 or 3 denotes a dependent ambulator who requires assistance from another person in the form of continuous manual contact (1), continuous or intermittent manual contact (2), or verbal supervision/guarding (3).
  A score of 4 or 5 describes an independent ambulator who can walk freely on: level surfaces only (4) or any surface (5=maximum score).
10 Meter Walk Test (10mWT) | Change from Baseline 10MWT at 4, 8 and 16 weeks
  The 10mWT is used to assess walking speed in meters/second (m/s) over a short distance. The total time taken to ambulate 6 meters (m) is recorded to the nearest hundredth of a second. 6 m is then divided by the total time (in seconds) taken to ambulate and recorded in m/s.
  The time is measured for the middle 6 m to allow for patient acceleration and deceleration.
  The time is started when any part of the leading foot crosses the plane of the 2-m mark.
  The time is stopped when any part of the leading foot crosses the plane of the 8-m mark.1 The time to walk the middle 6m, the level of assistance, and type of assistive device and/or bracing used will be documented.
  If a patient requires total assistance or is unable to ambulate at all, a score of 0 m/s will be documented.
Six-minute walk test (6MWT) | Change from Baseline 6MWT at 4, 8 and 16 weeks
  The 6MWT is a sub-maximal exercise test used to assess walking endurance and aerobic capacity. Participants will walk around the perimeter of a set circuit for a total of six minutes. The score of the test is the distance a patient walks in 6 minutes (measured in meters and can round to the nearest decimal point).
  Distance (in meters) covered in six minutes is calculated by multiplying the number of total laps by 12 meters and adding the distance of the partial lap completed at the time the test ended.
modified Barthel Index (mBI) | Change from Baseline mBI at 4, 8 and 16 weeks
  mBI for activities of daily living is meant to be used in the assessment of patient performance (or degree of assistance required) with respect to self-care, sphincter management, transfers and locomotion. The index consist of 10 items (each scored with a number of points) that relate to activities of daily living (ADLs) where the final score is calculated by summing the points awarded to each item. A five-point rating scales for each item to improve sensitivity to detecting change.
  The 10 items assessed relate to:
  * Help needed with feeding;
  * Help needed with bathing;
  * Help needed with grooming;
  * Help needed with dressing;
  * Presence or absence of fecal incontinence;
  * Presence or absence of urinary incontinence;
  * Help needed with transfers;
  * Help needed with walking;
  * Help needed with climbing stairs.
  Interpretation:
  * 91-100 Slight dependency
  * 61-90 Moderate dependency
  * 21-60 Severe dependency
  * 0-20 Total dependency
EuroQol- 5 Dimension (EQ-5D) | Change from Baseline EQ-5D at 4, 8 and 16 weeks
  EQ-5D is an instrument which evaluates the generic quality of life. The EQ-5D descriptive system is a preference-based HRQL measure with one question for each of the five dimensions that include mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The answers given to ED-5D permit to find 243 unique health states or can be converted into EQ- 5D index an utility scores anchored at 0 for death and 1 for perfect health.
Frontal Assessment Battery (FAB) | Change from Baseline FAB at 4, 8 and 16 weeks
  The FAB is a brief tool that can be used at the bedside or in a clinic setting to assist in discriminating between dementias with a frontal dysexecutive phenotype and Dementia of Alzheimer"s Type (DAT).
  The FAB has validity in distinguishing Fronto-temporal type dementia from DAT in mildly demented patients (MMSE > 24). Total score is from a maximum of 18, higher scores indicating better performance.
Stroop Colour Word Test (SCWT) | Change from Baseline SCWT at 4, 8 and 16 weeks
  The SCWT is a neuropsychological test extensively used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the simultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. The subject is asked to read the words in the first task, to name colors in the second and third tasks. It is necessary to mark both any mistakes made but also the time spent on each task. The cut-off for the error interference effect is 4.24, while the cut-off for the time interference effect is 36.92.
Digit Cancellation Test (DCT) | Change from Baseline DCT at 4, 8 and 16 weeks
  In the DCT the patient is asked to cross out with a pencil, as quickly as possible, all numbers corresponding to those indicated at the top of each matrix. Line A serves as an example. The performance of the subject is counted from line I. Corrections of the barriers are not allowed. The task of the examiner is mark the point at which the subject has exceeded the maximum time of the test, but let the subject let the subject finish his task for each matrix. The maximum time for each matrix is 45 sec- and is considered from the moment the subject finishes the run in. If the subject takes less time than the maximum time, it will be indicated at the end of each matrix. The time cut-off for the test is 23.9.
Trial Making Test (TMT) | Change from Baseline TMT at 4, 8 and 16 weeks
  The TMT measures flexibility of thinking on a visual-motor sequencing task. It consists of two parts, A and B, where 25 circles distributed over a sheet of paper. In Part A, the circles are numbered 1 - 25, and the patient should draw lines to connect the numbers in ascending order. In Part B, the circles include both numbers (1 - 13) and letters (A - L); as in Part A, the patient draws lines to connect the circles in an ascending pattern, but with the added task of alternating between the numbers and letters (i.e., 1-A-2-B-3-C, etc.).
  Results for both TMT A and B are reported as the number of seconds required to complete the task; therefore, higher scores reveal greater impairment.
  Trail A: Average 29 seconds, Deficient > 78 seconds, Rule of Thumb Most in 90 seconds Trail B: Average 75 seconds, Deficient > 273 seconds, Rule of Thumb Most in 3 minutes
Dual-Energy X-ray Absorptiometry (DEXA) | Change from Baseline DEXA at 4, 8 and 16 weeks
  DEXA is an instrumental examination based on the principle of differential attenuation of an X-ray beam, at two energy levels, as it passes through tissues. This attenuation is recordable and correlated with the body composition of the subject being examined.
  The device uses a coincident X-ray beam with no scattering in the environment. The radiation dose per single examination is minimal (1 mRem). There is therefore no risk to both patient and operator, and it is possible to repeat the examination at short intervals.
  DEXA allows for:
  1. a weight and percentage assessment of lean mass and fat mass in different body districts. It is therefore possible to determine the areas of fat accumulation and quantify their weight in grams.
  2. a selective assessment in the different body districts of the state of bone mineralization.
  The examination has a total duration of 30 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Giovannini, MD, phD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy